CLINICAL TRIAL: NCT05767593
Title: Clinical Validation of Samsung Smartwatch
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Amanda W. Baker, Ph.D., Director, Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital
Other Study IDs: 2022P002104
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder; Mood Disorders; Mental Health Issue
Keywords: Wearable technology; Smartwatch
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Depressed Adults: Adults with a current diagnosis of Major Depressive Episode
  Interventions: Device: Wearing Samsung smartwatch and filling out daily surveys
- Healthy Controls: Adults without a current or past diagnosis of Major Depressive Episode
  Interventions: Device: Wearing Samsung smartwatch and filling out daily surveys

INTERVENTIONS:
Device: Wearing Samsung smartwatch and filling out daily surveys — Participants will wear a Samsung smartwatch and fill out daily surveys about their mood and depressive symptoms.

SUMMARY:
Objective:

Wearable technology holds promising potential for mental health monitoring and detection. Samsung has developed an algorithm that they believe can detect signs of depression and anxiety in smartwatch users. They have used this algorithm to create a "Mindfulness Index," which is an easily understood visual index of mental health. The primary aim of the study is to evaluate the performance of Samsung's Mindfulness Index in identifying those who have received a diagnosis of Major Depressive Disorder (MDD) from a clinician-administered semi-structured diagnostic interview.

Research Procedures:

The target sample size is 135 individuals diagnosed with current Major Depressive Disorder and 85 healthy controls. To meet this target, the recruitment target is set at 220 participants. Participants will be assigned to the MDD condition, or the healthy control condition based on their score on the Beck Depression Inventory. Each subject will be followed for 3 months. Participants will be provided with a Samsung smartphone and Samsung smartwatch. Participants will be asked to wear the smartwatch 24 hours per day, except while charging. This smartwatch will collect data on heartrate, sleep time, and step count. During the study, each day participants will receive texts prompting a link to a "daily diary." These surveys will ask about depression and anxiety symptoms. Additionally, during the first 3 weeks of the study, participants will participate in ecological momentary assessment; texts will be sent 5 times per day prompting participants to fill out a survey about how they currently feel in that moment. These extra surveys will stop after the first 3 weeks of the study, but the daily diary surveys will continue throughout the study. Furthermore, virtual clinician visits will occur at weeks 4, 8, and 12.

ELIGIBILITY:
Inclusion Criteria (Depressed Adults)

1. Age 18-65
2. Meet full DSM-5 diagnostic criteria for a current major depressive episode, as assessed by the MINI for DSM-5 or Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) AND exhibit both:

   1. Beck Depression Inventory score of 9 or higher.
   2. Clinical Global Impressions Scale of 3 or higher.
3. If the patient is receiving psychopharmacological or psychosocial treatment, must be stable for 8 weeks prior to enrollment.

Inclusion Criteria (Healthy Controls)

1. Age 18-65
2. Do not meet the criteria for current or past major depressive episodes according to the DSM-5 criteria AND exhibit both:

   1. Beck Depression Inventory score of 8 or lower.
   2. Clinical Global Impressions Scale of 2 or lower.
3. If the patient is receiving psychopharmacological or psychosocial treatment, must be stable for 8 weeks prior to enrollment.

Exclusion Criteria

1. A lifetime history of bipolar disorder, schizophrenia, psychosis, or delusional disorders; an eating disorder in the past 6 months; organic brain syndrome; a history of substance use disorder in the last 12 months.
2. Presence or history of clinically significant neurological disorders and brain injuries (cerebral infarction, cerebral hemorrhage, multiple sclerosis, epilepsy, etc.)
3. Serious medical illness or instability for which hospitalization may be likely within the next year.
4. Patient does not own a smartphone with a data plan that allows them to receive text messages and access the internet throughout the day.
5. Patient is unable to understand study procedures and participate in the informed consent process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: U.S. residents recruited through online advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Performance of an index derived from passively collected data in identifying those who have received a diagnosis of Major Depressive Disorder (MDD) | Up to 3-months
  Area under the Receiver-Operating Characteristic curve (AUC) for an index derived from up to 3-months of passively-collected data from a smartwatch device in identifying those diagnosed with major depressive disorder (as assessed by MINI or DIAMOND Diagnostic Interview).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Baker, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Anxiety and Traumatic Stress Disorders, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No